CLINICAL TRIAL: NCT00678275
Title: Prophylaxis of Chronic Graft-versus-host Disease (cGvHD) With or Without Anti-T-lymphocyte-globulin (ATG Fresenius) Prior Allogeneic Peripheral Stem Cell Transplantation From HLA-identical Siblings After Myeloablative Conditioning in Patients With Acute Leukemia: A Randomized Phase III-study
Brief Title: Chronic Graft-versus-host Disease (cGvHD) Prophylaxis With or Without ATG Prior to Stem Cell Transplantation (SCT) From HLA-identical Siblings in Patients With Acute Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATGFamilyStudy
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Hematopoeitic Stem Cell Transplantation from HLA-identical sibling, RECEIVING ATG in conditioning regimen
  Interventions: Drug: ATG FRESENIUS (Anti-Lymphocyte-Globulin)
- B (Other): Hematopoeitic Stem Cell Transplantation from HLA-identical sibling, NOT RECEIVING ATG in conditioning regimen
  Interventions: Drug: ATG FRESENIUS (Anti-Lymphocyte-Globulin)

INTERVENTIONS:
Drug: ATG FRESENIUS (Anti-Lymphocyte-Globulin) — conditioning regimen with ATG: ATG FRESENIUS dosing: 10mg/kg/day, (day -3, -2,-1) when randomised Arm A
  Arms: A
Drug: ATG FRESENIUS (Anti-Lymphocyte-Globulin) — conditioning regimen WITHOUT ATG when randomised Arm B
  Arms: B

SUMMARY:
This multicenter, prospective phase III-study is to compare the administration of ATG FRESENIUS to the NON-administration of ATG FRESENIUS in a myeloablative conditioning regimen followed by allogeneic hematopoeitic stem cell transplantation from an HLA-identical sibling in patients with acute Leukemia. This clinical trial is to show that the administration of ATG FRESENIUS reduces the risk of chronic Graft-versus-Host disease after allogeneic stem cell transplantation from HLA-identical siblings.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia in first or subsequent complete remission (de-novo or secondary AML)
* Acute lymphoblastic leukemia in first or subsequent complete remission
* Patient's age: 18 - 65 years
* Myeloablative standard conditioning
* HLA-identical sibling (HLA-A, HLA-B, HLA-DRB1 and HLA-DQB1)
* No major organ dysfunctions
* Patient's written consent

Exclusion Criteria:

* No complete remission at time of randomization
* Severe irreversible renal, hepatic, pulmonary or cardiac disease, such as

  * Total bilirubin, SGPT or SGOT 5 times upper the normal level
  * left ventricular ejection fraction <30%
  * Creatinine clearance <30 ml/min
  * DLCO <35% and/or receiving supplementary continuous oxygen
* Positive serology for HIV
* Pregnant or lactating women
* Serious psychiatric or psychological disorders
* Progressive invasive fungal infection at time of registration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2006-10; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
comparison of cumulative incidence of chronic GvHD (limited or extensive) after allogeneic SCT from HLA-identical siblings with or without anti-T-lymphocyte-globulin at 2 years after transplantation | 2 years after transplantation

SECONDARY OUTCOMES:
comparison of: acute GvHD/quality of life/treatment-related mortality/toxicity/ overall survival/progression-free survival/engraftment/chronic-GvHD-free survival | 2 years after transplantation
incidence of infection/ AEs and ADRs | 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department for Stem Cell Transplantation
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Chakupurakal G, Freudenberger P, Skoetz N, Ahr H, Theurich S. Polyclonal anti-thymocyte globulins for the prophylaxis of graft-versus-host disease after allogeneic stem cell or bone marrow transplantation in adults. Cochrane Database Syst Rev. 2023 Jun 21;6(6):CD009159. doi: 10.1002/14651858.CD009159.pub3. PMID 37341189
- [Derived] Bonifazi F, Solano C, Wolschke C, Sessa M, Patriarca F, Zallio F, Nagler A, Selleri C, Risitano AM, Messina G, Bethge W, Herrera P, Sureda A, Carella AM, Cimminiello M, Guidi S, Finke J, Sorasio R, Ferra C, Sierra J, Russo D, Benedetti E, Milone G, Benedetti F, Heinzelmann M, Pastore D, Jurado M, Terruzzi E, Narni F, Volp A, Ayuk F, Ruutu T, Kroger N. Acute GVHD prophylaxis plus ATLG after myeloablative allogeneic haemopoietic peripheral blood stem-cell transplantation from HLA-identical siblings in patients with acute myeloid leukaemia in remission: final results of quality of life and long-term outcome analysis of a phase 3 randomised study. Lancet Haematol. 2019 Feb;6(2):e89-e99. doi: 10.1016/S2352-3026(18)30214-X. PMID 30709437
- [Derived] Kroger N, Solano C, Wolschke C, Bandini G, Patriarca F, Pini M, Nagler A, Selleri C, Risitano A, Messina G, Bethge W, Perez de Oteiza J, Duarte R, Carella AM, Cimminiello M, Guidi S, Finke J, Mordini N, Ferra C, Sierra J, Russo D, Petrini M, Milone G, Benedetti F, Heinzelmann M, Pastore D, Jurado M, Terruzzi E, Narni F, Volp A, Ayuk F, Ruutu T, Bonifazi F. Antilymphocyte Globulin for Prevention of Chronic Graft-versus-Host Disease. N Engl J Med. 2016 Jan 7;374(1):43-53. doi: 10.1056/NEJMoa1506002. PMID 26735993